CLINICAL TRIAL: NCT05586659
Title: Epidemiology of Triple Negative Breast Cancer in Asyut Clinical Oncology Department From 2015 to 2022 ( A Hospital Based Study)
Brief Title: Epidemiology of TNBC in Asyut Clinical Oncology Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Saber Khalifa Mohammed, Doctor, Assiut University
Other Study IDs: TNBC
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiological Study about behavior of TNBC in Clinical oncology department in 8 y in Asyut university hospital

DETAILED DESCRIPTION:
Breast Cancer )BC) is the most Common malignancy in women in 2020, there were 2.3 million women diagnosed with breast cancer and 685.000 deaths globally. Breast cancer rates are 88% higher in developed countries compared to developing countries .

TNBC represents accounts for approximately 24% of all breast cancer in 2020 .While in Egypt it accounts for 11.05% according to Egyptian national BC (5). By gene expression profiling ,4 subtypes of TNBC emerged : luminal androgen receptor (LAR), mesenchymal stem-like (MSL), immunomodulatory (IM), basal-like (BL1 and BL2) . Most of cases are advanced with median survival about 14 months . Brain and visceral organs represent common sites of distant metastasis . So it is considered the worst prognosis . In addition , chemotherapy is only option in treatment with no available targeted options for decades. Now we have Immunotherapy (IO ) and PARP inhibitors in neoadjuvant (NAT) and metastatic setting For example : Key note 355 which add Pembrolizumab in NAT which lead to marked improvement in pathological complete response ( PCR ) And in high risk patient and have marked results in disease and event free survival(8) .Poly (ADP-ribase) poly merase -1 (PARP-1) inhibitors appear to particularly effective in BRCA 1/2 mutation carries (9) .As reviewed by rodleret al. emerging data suggest that BRCA 1/2 carriers with TNBC disease may respond favorably to cisplatin therapy .

ELIGIBILITY:
Inclusion Criteria:- Age ≥ 18

* Male or female
* Diagnosed as TNBC from ( 2015- 2022 ) confirmed by pathology
* Adjuvant or metastatic

Exclusion Criteria:- Have other type of malignancy

* HER2 , ER, PR positive

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: male or female with triple negative breast cancer Diagnosed as TNBC from ( 2015- 2022 ) confirmed by pathology
  - Adjuvant or metastatic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of TNBC | Baseline
  Incidence of TNBC in clinical oncology department from 2015-2022
Behavior of the disease and stage | baseline
  Behavior of the disease and stage of presentation
Types of treatment | baseline
  Types of treatment

SECONDARY OUTCOMES:
DFS | Baseline
  Disease free survival
PFS | Baseline
  progression free survival
OS | Baseline
  overall survival

REFERENCES:
- [Background] Wolff AC, Hammond ME, Hicks DG, Dowsett M, McShane LM, Allison KH, Allred DC, Bartlett JM, Bilous M, Fitzgibbons P, Hanna W, Jenkins RB, Mangu PB, Paik S, Perez EA, Press MF, Spears PA, Vance GH, Viale G, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. Recommendations for human epidermal growth factor receptor 2 testing in breast cancer: American Society of Clinical Oncology/College of American Pathologists clinical practice guideline update. J Clin Oncol. 2013 Nov 1;31(31):3997-4013. doi: 10.1200/JCO.2013.50.9984. Epub 2013 Oct 7. PMID 24101045
- [Background] Lin NU, Claus E, Sohl J, Razzak AR, Arnaout A, Winer EP. Sites of distant recurrence and clinical outcomes in patients with metastatic triple-negative breast cancer: high incidence of central nervous system metastases. Cancer. 2008 Nov 15;113(10):2638-45. doi: 10.1002/cncr.23930. PMID 18833576